CLINICAL TRIAL: NCT04104555
Title: Orthotics for Treatment of Symptomatic Flat Feet in Children the OSTRICH Study
Brief Title: Orthotics for Treatment of Symptomatic Flat Feet in Children
Acronym: OSTRICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of York (Other)
Collaborators: University of Leeds (Other); University of Salford (Other); University of Oxford (Other); King's College London (Other); University of Warwick (Other)
Responsible Party: Principal Investigator, Sarah Cockayne, Research Fellow, University of York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 265719
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pes Planus
Keywords: Pes planus; Randomised controlled trial; Orthoses; Exercise; Children
MeSH Terms: conditions — Flatfoot; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Usual supportive care - exercises and footwear advice (Active Comparator): OSTRICH main trial:
  Participants will be offered an exercise programme and advice regarding footwear. The treating clinician will be able to prescribe appropriate exercises from a menu of exercises.
  Interventions: Other: Usual supportive care - exercises and footwear advice (the comparator)
- Prefabricated, off-the-shelf orthoses (Experimental): OSTRICH main trial:
  A pair of prefabricated, off-the-shelf orthoses (i.e. mass produced to a generic shape but can be adapted by a clinician) plus an exercise programme and advice regarding footwear. The treating clinician will be able to prescribe appropriate exercises from a menu of exercises.
  Interventions: Device: Prefabricated orthoses
- Signposting to multimedia (Experimental): OSTRICH 'signposting to multimedia' Study within a trial (SWAT) Participants will be given signposting information to the multimedia trial information resources in the participant information sheet which is included in the OSTRICH recruitment pack.
  Interventions: Other: Signposting to multimedia
- Standard written information only (No Intervention): OSTRICH signposting to multimedia' Study within a trial (SWAT) Participants will receive the standard written information sheet only. This will not include signposting to the multimedia trial information resources, in the OSTRICH recruitment pack.
- Birthday card (Experimental): OSTRICH Birthday card study within a trial (SWAT) Participants will be sent a birthday card on or shortly before their birthday from the OSTRICH study team to encourage completion of questionnaires.
  Interventions: Other: Birthday card
- No birthday card (No Intervention): OSTRICH Birthday card study within a trial (SWAT) Participants will not be sent a birthday card during the trial.

INTERVENTIONS:
Other: Birthday card — Birthday card sent to participants in the post
  Arms: Birthday card
Device: Prefabricated orthoses — Prefabricated insole
  Arms: Prefabricated, off-the-shelf orthoses
Other: Signposting to multimedia — Signposting to multimedia information in the patient information sheet which is sent to participants in the post as part of the OSTRICH recruitment pack.
  Arms: Signposting to multimedia
Other: Usual supportive care - exercises and footwear advice (the comparator) — Active comparator
  Arms: Usual supportive care - exercises and footwear advice

SUMMARY:
Update 13.12.2021 To mitigate the effects the COVID-19 pandemic, and due to difficulties in sites setting up the custom orthoses arm of the protocol an amendment was approved to change the design of the study from a 3 to a 2 arm trial. The amendment drops the custom orthoses arm and was implemented prior to the start of recruitment.

As a child grows the shape of their foot changes and most develop an arch in their foot. For some, however, the arch does not fully form or it might be flat against the ground. This is known as having flat feet and it can cause pain in the feet, legs, or back. At the moment, we are not sure what the best treatment for flat feet is, so the purpose of this research is to conduct a trial to compare two of the most common treatments. The first is exercise and advice about things like which types of shoes might help. The second of the treatment is a type of insole, which is put inside the shoe.

Participants will receive their treatment as part of their normal National Health System care. We would like 478 children and young people aged between 6 and 14 years old to take part in the study. Everyone will receive advice about the type of shoes to wear, ankle exercises and things to look out for when children have painful flat feet. In addition to this, half of the participants will receive a pre-made insole that is the right size. We will ask for their help for 12 months. During this time, we will track their progress by sending them 3 questionnaires in the post to fill in and weekly text messages to find out how painful their feet are during the first few months. We also want to learn more about the problems that flat feet cause, and children's experiences of the treatments delivered as part of this clinical trial. We will explore this through in-depth conversations with children and their parent(s) or the person who looks after them. Once we have finished the trial, we will work with the people who took part in the trial, and clinicians, to make sure that our results can be used by as many people as possible.

We will run 3 additional studies. The first will find out if having information about the study in the form of a video in addition to information in a paper booklet will increase recruitment rates. The second will find out if sending participants a birthday card will increase the response rates to postal questionnaires. The third study will take a 3D impression of the participant's foot and see if it changes over the course of the study.

DETAILED DESCRIPTION:
The aim of the study is to undertake a large, pragmatic, multi-armed, randomised controlled trial to assess the clinical and cost-effectiveness of prefabricated orthoses in addition to exercises and advice compared with exercises and advice alone on the physical functioning of children with symptomatic flat feet. We will aim to recruit 478 children with flat feet. They will be allocated to one of two groups, in a 1:1 ratio to either (a) prefabricated orthoses plus exercises and footwear advice or (b) exercises and footwear advice only. We will follow the participants up for 12 months after randomisation to assess their physical functioning, levels of pain and quality of life. We will undertake qualitative interviews with approximately 30 children and their parents, to find out about their experiences of having flat feet, and of being in the trial.

In addition to the main OSTRICH study we will undertake two additional trial methodological Studies within a Trial (SWAT) and a sub-study.

The multimedia trial information SWAT: This SWAT will evaluate the effectiveness of including signposting to multimedia trial information in the patient information sheet, which is sent to participants in their recruitment pack.

The birthday card SWAT: This SWAT will evaluate the effectiveness of sending a birthday card to participants on response rates to postal questionnaires.

Foot scan sub-study: This embedded observational sub-study will assess the capability of a 3D scanning approach to identify and stratify severity of pes planus and to assess change in foot shape over the duration of the trial. We will investigate the associations between aspects of foot shape and score on the physical domain scale of the OxAFQ-C.

ELIGIBILITY:
OSTRICH main trial inclusion criteria:

Potential participants will be included in the trial if they fulfil all of the following criteria:

* Are aged between six and 14 years, inclusive
* Have one or both symptomatic pes planus*
* The child and/or parent/legal guardian is able to speak, write and understand English
* The parent/legal guardian is able to give informed consent *Symptomatic pes planus is described as the manifestation of foot and lower limb symptoms, secondary to altered foot alignment (reduced medial longitudinal arch, everted rearfoot and abducted forefoot). The diagnosis will be made pragmatically, by treating clinicians in line with current practice

OSTRICH main trial exclusion criteria:

Potential participants will be excluded from the study if they fulfil any of the following criteria:

* Have a history of major trauma or fracture of the lower leg (below knee)
* Have pes planus secondary to any systematic condition/syndrome** /malignancy
* Have a history of foot and/or ankle surgery
* Require an ankle-foot orthoses or other lower limb device or have received treatment previously for their flat feet

  * This does not exclude children with hypermobility spectrum disorder (HSD) where the manifestation is non-syndromic and isolated (L-HSD), peripheral (P-HSD) or generalised hypermobility (G-HSD)(14).

OSTRICH signposting to multimedia trial information SWAT: inclusion criteria any potential participant identified as eligible to be sent trial information from a site taking part in the SWAT, will be eligible for the study.

OSTRICH birthday card SWAT Inclusion criteria: All participants recruited into the host trial will be eligible to take part in this SWAT. Exclusion criteria: Any participant who has withdrawn from the main OSTRICH study or is not due a follow up questionnaire will be excluded.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Physical domain subscale of the Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) over the 12 month follow-up period. | For the primary comparison the physical domain subscale will be compared between the groups using a linear covariance pattern mixed model to estimate the effect over the whole 12 month followup, incorporating data from all available time points
  The OxAFQ-C is a self-report health status measure questionnaire for child patients (aged 5-14) affected by foot and ankle conditions that are considered important to children. There are three domains, whose domain scores are reported separately (ie there is no total score). For the primary outcome however, we will just use the physical domain subscale. There are 6 items on the 'Physical' domain. The response options to each item are on a 5-point scale rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), where the number in brackets represents the value that should be applied to each response. The total 'physical domain score' is divided by the maximum for the domain ie 24. This score can then be transformed to a percentage scale (0-100) to aid interpretation. A higher score for a domain represents better functioning. This will be rated by the child (participant) and their parent/legal guardian using a proxy version.

SECONDARY OUTCOMES:
The 'School and Play' domain of the Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) | Collected at baseline, 3,6 and 12 months post randomisation
  The OxAFQ-C is a self-report health status measure questionnaire for child patients (aged 5-14) affected by foot and ankle conditions that are considered important to children. There are three domains, whose domain scores are reported separately (ie there is no total score). However for the secondary outcome we will use the 'School and Play' domain. There are 4 items on the 'School and Play' domain. The response options to each item are on a 5-point scale rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), where the number in brackets represents the value that should be applied to each response. The total of the 'School and Play' domain score is divided by the maximum for the domain ie 16. This score can then be transformed to a percentage scale (0-100) to aid interpretation. A higher score for a domain represents better functioning. This will be rated by the child (participant) and their parent/legal guardian using a proxy version.
The 'Emotional' subscale of the Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) | Collected at baseline, 3,6 and 12 months post randomisation
  The OxAFQ-C is a self-report health status measure questionnaire for child patients (aged 5-14) affected by foot and ankle conditions that are considered important to children.
  There are three domains, whose domain scores are reported separately (ie there is no total score). However for the secondary outcome we will use the 'Emotional' domain. There are 4 items on the 'Emotional' domain. The response options to each item are on a 5-point scale rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), where the number in brackets represents the value that should be applied to each response. The total of the 'Emotional' domain score is divided by the maximum for the domain score ie 16. This score can then be transformed to a percentage scale (0-100) to aid interpretation. A higher score for a domain represents better functioning. This will be rated by the child (participant) and their parent/legal guardian using a proxy version.
Footwear item of the Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) | Collected at baseline, 3, 6 and 12 months post randomisation
  The OxAFQ-C is a self-report health status measure questionnaire for child patients (aged 5-14) affected by foot and ankle conditions that are considered important to children. This item was added to reflect the concern by many children that they can or cannot wear the footwear they prefer. It is a 5-point scale rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), where the number in brackets represents the value. It is reported as a single item with higher score representing better functioning. This will be rated by the child (participant) and their parent/legal guardian using a proxy version.
EuroQoL-Five Dimension Youth | Collected at baseline, 3,6 and 12 months post randomisation
  The EuroQoL-5 Dimension Youth (EQ5DY) is a child friendly, generic quality of life measure. Health status is measured in terms of 5 domains: "mobility", "looking after myself", "doing usual activities", "having pain or discomfort" and "feeling worried, sad or unhappy". Each dimension has 3 levels ranging from 1 no problems, 2 some problems and 3 a lot of problems. The respondent is asked to indicate their health state by ticking in the box against the most appropriate statement in each of the 5 dimensions. From these 5 dimensions an EuroQoL-5 Dimension Youth (EQ5DY) value is calculated. This measure also includes a Visual Analogue Scale on how good or bad the participant's health is "today", on a vertical scale of 0 to 100. The endpoints of the scale are labelled "100 The best health you can imagine" and "0 The worst health you can imagine." This will be rated by the child (the participant) and their parent/legal guardian (using a proxy version).
Child Health Utility 9D (CHU9D) | Collected at baseline, 3,6 and 12 months post randomisation
  The Child Health Utility 9D (CHU9D) is a paediatric self-reported generic quality of life measure. It consists of nine dimensions; "worried", "sad", "pain", "tiredness" "annoyed", "school work/homework", "sleep", "daily routine" and "able to join in activities". The measure is rated on a five point scale on which the participants rate the level to how they are feeling, with a "don't" sentence linked with no problems (e.g. I don't feel sad today) and "very" with the participant experiencing a lot of problems (e.g. I feel very sad). Calculation of an universal score is supported by a specific scoring algorithm, with 1 representing 'full health' and 0 'death'. In this study the CHU9D is rated by the child (the participant) and their parent/legal guardian (using a proxy version).
Foot pain score measured by numeric rating scale | Collected once a week for 12 weeks and at baseline, 3, 6 and 12 months post randomisation
  Self-report pain status will be measured using a Numeric Rating Scale (NRS) of 0 to 9. The participant will be asked to estimate their pain intensity over the past week, where 0 indicates no pain at all and 9 the worst pain. In this study the foot pain score with numeric rating is rated by the participant's parent/legal guardian .
Healthcare resource use | Collected at baseline, 3,6 and 12 months post randomisation
  Self report healthcare resource use. Healthcare utilisation will be recorded in primary care and the community and within the hospital setting.
Foot pain over past week measured by Wong-Baker Faces pain rating scale | Collected at baseline, 3,6 and 12 months post randomisation
  Self-report measure of pain in left and right feet, using Wong-Baker faces pain rating scale (0-10) where 0 indicates no pain at all and 10 being the worst possible pain. In this study the foot pain score is rated by the child (the participant).

OTHER OUTCOMES:
Proportion of participants who go on to be randomised to the OSTRICH trial. | Post randomisation
  Primary outcome for the 'pen and signposting to multimedia trial information Study within a Trial
Retention to main OSTRICH trial | 3, 6 and 12 months post randomisation
  Secondary outcome for the 'pen and signposting to multimedia trial information Study within a trial
Response rate to the participant follow-up questionnaire at the first time point following receipt of the birthday card | Next followup either , 3, 6 or 12 months post randomisation
  Primary outcome to 'birthday card' Study within a Trial
Response rate to the participant follow-up paper questionnaire at the 12-month follow-up | 12 months post randomisation
  Secondary outcome to 'birthday card' Study within a Trial
Completeness of host-trial primary outcome measure | 12 months post randomisation
  Secondary outcome to 'birthday card' Study within a Trial
Time to return postal questionnaire | 3, 6 and 12 months post randomisation
  Secondary outcome to 'birthday card' Study within a Trial
Need for questionnaire reminder | 3, 6 and 12 months post randomisation
  Secondary outcome to 'birthday card' Study within a Trial
Qualitative interviews | Interviews will be conducted throughout the study
  Parental/legal guardian and child experiences and management of pes planus
3D foot scan | Baseline and at 12 months
  3D scan of both feet

CONTACTS AND LOCATIONS:
Overall Officials: David Torgerson, PhD, Principal Investigator — University of York
Locations (16):
- United Kingdom (16):
  - East Cheshire NHS Trust, Macclesfield, Cheshire
  - Birmingham Community Healthcare NHS Foundation Trust, Birmingham
  - Bolton NHS Foundation Trust, Bolton
  - Cardiff and Vale University Local Health Board, Cardiff
  - Medway Community Healthcare, Gillingham
  - North Lincolnshire & Goole NHS Foundation Trust, Goole
  - Harrogate and District Foundation Trust, Harrogate
  - Leeds Community Healthcare NHS Trust, Leeds
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Kent Community Health NHS Foundation Trust, Maidstone
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Lancashire & South Cumbria Nhs Foundation Trust, Preston
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Solent NHS Trust, Southampton
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore
  - Walsall Healthcare NHS Trust, Walsall

IPD SHARING:
Plan to Share IPD: No
Requests for OSTRICH study data may be submitted to the Chief Investigator once the results of the study have been published. Requests will be dealt with on a case by case basis and in accordance with the University of York, Department of Health Sciences, York Trials Unit's Standard Operating Procedures.

REFERENCES:
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub4. PMID 35080267
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 14;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub3. PMID 35029841